CLINICAL TRIAL: NCT05481203
Title: The Effect Of Distraction Methods On Fear And Anxiety In Children Before The Covid 19 Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hatice Uzşen, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Distraction
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Anxiety; Fear
Keywords: COVID-19 test; nasopharyngeal swab collection; pediatric nursing; distraction methods
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This was an RCT with parallel groups conducted between March, 2022 and August, 2022 at the pediatric emergency unit of a hospital in Black Sea Region Turkey
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Kaleidescope Group (Experimental): Kaleidoscope Group: it and asking about the colors and shapes seen within it. This distraction procedure started before the procedure and continued until it ended.
  Interventions: Behavioral: The Kaleidescope
- The Visual Illusion Cards Group (Experimental): The Visual Illusion Cards Group: Just before the nasopharyngeal swab participants were allowed to check the cards and were asked what they saw in them.
  Interventions: Behavioral: The visual illusion cards
- The Control Group (No Intervention): The control group received the routine nasopharyngeal swab procedure and did not receive any other nonpharmacological intervention

INTERVENTIONS:
Behavioral: The Kaleidescope — During the nasopharyngeal swab collection process, the researcher held a kaleidoscope to each child's eye, leisurely turning it and asking about the colors and shapes seen within it.
  Arms: The Kaleidescope Group
Behavioral: The visual illusion cards — Just before the nasopharyngeal swab participants were allowed to check the cards andwere askedwhat they saw in them.
  Arms: The Visual Illusion Cards Group

SUMMARY:
Aim: This research will be carried out to determine the effect of distracting methods on fear and anxiety in children before the COVID test.

DETAILED DESCRIPTION:
Inroduction: In the literature review, it has been seen that the positive effect of different nanpharmacological methods is supported to reduce pain and anxiety caused by medical procedures. Non-pharmacological methods are classified as physical methods, cognitive behavioral methods, and environmental or emotional intervention methods. In order to draw attention to another direction, which is among these methods; watching cartoons, inflating balloons, creating balloons by blowing foam, talking about things unrelated to the initiative, virtual reality glasses, listening to music, using kaleidoscope and distraction cards etc. is located. The subject of the study is the application of distraction methods in reducing the pain associated with short-term medical interventions.

ELIGIBILITY:
Inclusion Criteria:

* children who will be taken samples for Covid 19 test
* being between the ages of 5 to 10 years,
* literate

Exclusion Criteria:

* having chronic diseasesvisual
* audio, or speech impairments
* mental disorders,
* history of sedative, analgesic, or narcotic use within 24 h before admission
* inflammatory disease during admission.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
changing the anxiety in the Kaleidoscope group | up to 6 months
  changing the anxiety scores of the children in the Kaleidoscope group during Covid 19 test
changing the fear in the Kaleidoscope group | up to 6 months
  changing the fear scores of the children in the Kaleidoscope group during Covid 19 test
changing the anxiety in the Visual Illusion Cards group | up to 6 months
  changing the anxiety scores of the children in the Visual Illusion Cards group during Covid 19 test
changing the fear in the Visual Illusion Cards group | up to 6 months
  changing thefear scores of the children in the Visual Illusion Cards group during Covid 19 test

SECONDARY OUTCOMES:
changing the "Child Anxiety Scale-Stateness" score | up to 6 months
  The Children's Anxiety Meter (CAM) used. It assesses children's anxiety in clinical settings and uses before medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom, also includes horizontal lines at intervals going up to the top. Children are asked to mark how he/she feel "right now" to measure state anxiety. Scores range from 0 to 10.
changing the "Child Fear Scale" score | up to 6 months
  The Child Fear Scale (CFS) used. This one-item scale consists of five sex-neutral faces. It ranges from a no fear (neutral) face on the far left to a face showing extreme fear on the far right. The rater responds indicates the level of fear. Scores range from 0 to 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No